CLINICAL TRIAL: NCT00347984
Title: The Effect of Systane® Compared to Marketed Artificial Tears on Frequency of Drop Use
Brief Title: Product Preference With Systane Compared to Artificial Tears on Frequency of Drop Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: ORA, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 05-004-09
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2008-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Other: Systane Lubricant eye drops

SUMMARY:
The objective of this study was to evaluate the effect of Systane® compared to marketed artificial tears on the frequency of drop use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 (minimum); reported history of dry eye syndrome in both eyes; TFBUT ≤ 7 seconds in at least 1 eye at Visit 1; ≥ 1+ fluorescein staining score in any region in at least 1 eye at Visit 1; desire to use an artificial tear substitute for dry eye symptoms at least 4 times per day at Visit 1 and Visit 2.

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-12; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Frequency of drop use and/or desire to use; Drop preference

SECONDARY OUTCOMES:
Product questionnaire; Symptoms; Corneal and conjunctival staining; Tear film break-up time (TFBUT).

CONTACTS AND LOCATIONS:
Overall Officials: Mike Christensen, Study Director — Alcon Research
Locations (1):
- Maryland, Andover, Massachusetts, United States